CLINICAL TRIAL: NCT05641571
Title: Effects of an Exercise Intervention on Taxane-induced Peripheral Neuropathy in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CF22200A
Record Dates: First submitted 2022-10-26; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: CIPN - Chemotherapy-Induced Peripheral Neuropathy
Keywords: Taxane-induced peripheral neuropathy, extremity exercise

STUDY DESIGN:
Intervention Model Description: The 3~6 months home-based extremity exercise program will be intervened between newly diagnosed with breast cancer to the completion of chemotherapy. Participants have to perform a total of 50 minutes of exercise including the Ten Skilled Hand exercise fourth a day, 5 minutes each time and Buerger Allen exercise twice a day, 15 minutes each time. The observational group will need to record the extra exercise performed and the exercise prescription will be distributed after the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The 3~6 months home-based extremity exercise program will be intervened between newly diagnosed with breast cancer to the completion of chemotherapy. Participants have to perform a total of 50 minutes of exercise including the Ten Skilled Hand exercise fourth a day, 5 minutes each time and Buerger Allen exercise twice a day, 15 minutes each time.
  Interventions: Behavioral: The home-based extremity exercise program
- Observational group (No Intervention): The observational group will need to record the extra exercise performed and the exercise prescription will be distributed after the study.

INTERVENTIONS:
Behavioral: The home-based extremity exercise program — Participants have to perform a total of 50 minutes of exercise including the Ten Skilled Hand exercise fourth a day, 5 minutes each time and Buerger Allen exercise twice a day, 15 minutes each time before chemotherapy to the completion of chemotherapy.
  Arms: Exercise group

SUMMARY:
The purpose of this study is to examine the effects of an exercise program on the management of TIPN in breast cancer survivors. This experimental study utilizes purposive sampling to recruit 88 adults, newly diagnosed with stage I~III breast cancer women, who are expected to be treated with Taxane chemotherapy in a medical center located in central Taiwan. Participants will be randomly allocated to the experimental or observational group. The main outcomes are peripheral neuropathy and neuropathic pain. The 3~6 months home-based extremity exercise program will be intervened between newly diagnosed with breast cancer to the completion of chemotherapy. Participants have to perform a total of 50 minutes of exercise including the Ten Skilled Hand exercise fourth a day, 5 minutes each time and Buerger Allen exercise twice a day, 15 minutes each time. This study expects that the extremity exercise program will be able to prevent and manage peripheral neuropathy and neuropathic pain via increasing blood circulation. Moreover, the exercise program may also improve functioning and QOL in breast cancer survivors receiving Taxane chemotherapy.

DETAILED DESCRIPTION:
The incidence of breast cancer increases yearly. Taxane is one of the main chemotherapy drugs for breast cancer treatment. Taxane-induced peripheral neuropathy (TIPN) impairs breast cancer survivors' functioning, increases the risk of falls, and impacts quality of life (QOL). As TIPN worsens, there is a need to decrease chemotherapy dosage or terminate treatment. This may reduce the effect of chemotherapy, in addition, to increasing survivor's mortality. Up to date, no evidence-based, effective nonpharmacologic intervention to prevent or manage TIPN. Furthermore, no interventions were recommended by the U.S. Food and Drug Administration or TIPN expert organizations to prevent or treat TIPN. Therefore, the purpose of this study is to examine the effects of an exercise program on the management of TIPN in breast cancer survivors.

This experimental study utilizes purposive sampling to recruit 88 adults, newly diagnosed with stage I~III breast cancer women, who are expected to be treated with Taxane chemotherapy in a medical center located in central Taiwan. Participants will be randomly allocated to the experimental or observational group using the two strata: (1) adjuvant or neoadjuvant and (2) paclitaxel, docetaxel, or Taxane plus Platinum. Participants who have peripheral neuropathy before chemotherapy or regular exercise are excluded. The four-measure points are as the followings: (T1) before chemotherapy, (T2) after the completion of the first Taxane, (T3) the completion of half chemotherapy regimen, and (T4) the completion of chemotherapy. The main outcomes are peripheral neuropathy and neuropathic pain. The blood circulation of extremities, functional status, falls and QOL are also measured. SPSS 22 is used to enter and analyze data. Mean, standard deviation, frequency, and percentage are utilized to describe the distribution of the sample and research variables. Chi-squared and generalized estimating equation is used to detect the difference and change over time between the two groups.

The 3~6 months home-based extremity exercise program will be intervened between newly diagnosed with breast cancer to the completion of chemotherapy. Participants have to perform a total of 50 minutes of exercise including the Ten Skilled Hand exercise fourth a day, 5 minutes each time and Buerger Allen exercise twice a day, 15 minutes each time. The observational group will need to record the extra exercise performed and the exercise prescription will be distributed after the study. This study expects that the extremity exercise program will be able to prevent and manage peripheral neuropathy and neuropathic pain via increasing blood circulation. Moreover, the exercise program may also improve functioning and QOL in breast cancer survivors receiving Taxane chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be randomly allocated to the experimental or observational group using the two strata: (1) adjuvant or neoadjuvant and (2) paclitaxel, docetaxel, or Taxane plus Platinum.

Exclusion Criteria:

* Participants who have peripheral neuropathy before chemotherapy or regular exercise are excluded.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of peripheral neuropathy | Change of peripheral neuropathy from baseline measure at 6 months
  Total Neuropathy Score- clinical version, pain 0~100 Visual Analogue Scale, Identification Pain Questionnaire

SECONDARY OUTCOMES:
The score change in quality of life | Change of quality of life from baseline measure at 6 months
  Functional Assessment for Chronic disease Therapy- Taxane

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chiang Hung, Doctor, Principal Investigator — Taichung Veterans General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang YJ, Hung MC, Wu CJ, Huang CC, Cao HW. Effects of an exercise program on chemotherapy-induced peripheral neuropathy in newly diagnosed breast cancer individuals receiving taxanes: a randomized controlled trial. Support Care Cancer. 2025 Nov 10;33(12):1036. doi: 10.1007/s00520-025-10121-8. PMID 41212417